CLINICAL TRIAL: NCT07343479
Title: A Clinical Study of Sac-TMT for Injection Combined With Third-Generation Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) ± Radiotherapy in Subjects With EGFR-Mutated Non-Squamous Non-Small Cell Lung Cancer and Brain Metastasis Who Have Failed Prior EGFR-TKI Treatment
Brief Title: Sacituzumab Tirumotecan Plus Third-Generation TKI With/Without Radiotherapy for EGFR-Mutant NSCLC Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Fan Yun, MD, Director of the Department of Thoracic Oncology, Zhejiang Cancer Hospital, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2025-1523（IIT）
Record Dates: First submitted 2025-12-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); EGFR Gene Mutations; Brain Metastasis
Keywords: NSCLC with brain metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sac-TMT plus EGFR-TKI (Experimental): Sacituzumab tirumotecan combined with third-generation EGFR-TKI with or without intracranial radiotherapy
  Interventions: Drug: sac-TMT plus EGFR-TKI

INTERVENTIONS:
Drug: sac-TMT plus EGFR-TKI — Eligible subjects will receive sac-TMT (4 mg/kg, twice weekly (Q2W)) + third-generation EGFR-TKI ± intracranial radiotherapy. The decision to initiate intracranial radiotherapy will be determined by the investigator based on the patient's clinical condition.

SUMMARY:
This is a prospective, open-label, multi-center, single-arm clinical trial

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of sac-TMT combined with third-generation EGFR-TKI with/without intracranial radiotherapy in subjects with EGFR-mutated NSCLC and brain metastasis who have failed prior EGFR-TKI treatment. Eligible subjects will receive sac-TMT (4 mg/kg, twice weekly (Q2W)) + third-generation EGFR-TKI ± intracranial radiotherapy. The decision to initiate intracranial radiotherapy will be determined by the investigator based on the patient's clinical condition.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years at the time of signing the informed consent form (ICF), regardless of gender;
* Histologically or cytologically confirmed non-squamous NSCLC, and metastatic (Stage IV);
* Confirmed EGFR sensitizing mutation including exon 19 deletion (19-Del) or exon 21 point mutation (L858R);
* Subject has previously received EGFR-TKI therapy for locally advanced or metastatic disease and has experienced radiological PD;
* Subjects with new or previously diagnosed brain metastasis confirmed by contrast-enhanced cranial MRI;
* ECOG performance status scale of 0 or 1;
* Life expectancy ≥ 12 weeks;
* Adequate organ and bone marrow function;

Exclusion Criteria:

* Tumor histology or cytology confirms combined small cell lung cancer (SCLC), neuroendocrine carcinoma, carcinosarcoma components, or squamous cell carcinoma;
* Known leptomeningeal metastases;
* Other malignant tumors within 3 years prior to the first dose (except for tumors cured by local treatment, such as basal cell carcinoma of skin, squamous cell carcinoma of skin, cervical carcinoma in situ, etc.);
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, uncontrolled symptomatic arrhythmia, prolongation of QTcF interval to >470 ms, and other serious cardiovascular and cerebrovascular diseases within 6 months before study intervention;
* Uncontrolled systemic diseases as judged by the investigators;
* Clinically severe pulmonary impairment due to concurrent lung disorders, including but not limited to any underlying lung disorder (e.g., pulmonary embolism within 3 months before the first dose, severe asthma, severe chronic obstructive pulmonary disease, restrictive pulmonary disease, pleural effusion, etc.) or any autoimmune, connective tissue, or inflammatory disease that may involve the lungs (i.e., rheumatoid arthritis, sicca syndrome, sarcoidosis, etc.), or prior pneumonectomy;
* Subjects with active chronic inflammatory bowel disease, gastrointestinal obstruction, severe ulcer, gastrointestinal perforation, intra-abdominal abscess, or acute gastrointestinal hemorrhage;
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease;
* Active infection requiring systemic therapy;
* Active hepatitis B [hepatitis B surface antigen (HBsAg) positive, requiring hepatitis B virus deoxyribonucleic acid (HBV-DNA) testing; HBV-DNA ≥500 IU/mL or above the lower limit of detection, whichever is higher] or hepatitis C [hepatitis C antibody positive, and hepatitis C virus ribonucleic acid (HCV-RNA) above the lower limit of detection];
* Positive human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection;
* History of allogeneic tissue/solid organ transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-06-20 (Estimated); Study Completion 2029-12-20 (Estimated)

PRIMARY OUTCOMES:
6-month PFS rate | 6 months post treatment initiation date (maximum follow-up of 36 months)
  6-month PFS rate as assessed by the investigators according to RECIST v1.1.

SECONDARY OUTCOMES:
Overall ORR and DCR | From initiation of treatment to disease progression or death from any cause, whichever occurs first (maximum follow-up of 36 months)
  Overall ORR and DCR as assessed by the investigators according to RECIST v1.1
DOR | From first disease response until tumor progression (maximum follow-up of 36 months).
  DOR as assessed by the investigators according to RECIST v1.1
OS | From treatment initiation to death due to any cause or last day of contact, whichever occurred first (maximum follow-up of 36 months)
  Time from treatment initiation to date of death due to any cause or last day of contact.
Safety endpoints | From first dose of study treatment until 30 days after the last dose, assessed up to 36 months.
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) [based on the latest version of the Common Terminology Criteria for Adverse Events (CTCAE) of the National Cancer Institute (NCI)]

CONTACTS AND LOCATIONS:
Overall Officials: Yun Fan, Doctor, Study Director — Zhejiang Cancer Hospital; Hui Li, Doctor, Study Director — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No